CLINICAL TRIAL: NCT04159467
Title: Effect of Pelvic Floor Muscle Training on Urinary Incontinence Reports in Obese Women Undergoing a Low Calorie Diet Prior to Bariatric Surgery: an Assessor Blinded Randomized Controlled Trial
Brief Title: Effect of Pelvic Floor Muscle Training on Urinary Incontinence Reports in Obese Women Undergoing a Low Calorie Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Pauliana Carolina de Souza Mendes, Physiotherapist, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16379919.5.0000.5440
Record Dates: First submitted 2019-10-21; First posted 2019-11-12 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Urinary Incontinence; Obesity; Strength; Pelvic Floor
Keywords: Urinary Incontinence; Obesity; Diet; Pelvic floor muscles training
MeSH Terms: conditions — Urinary Incontinence; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator will be blind in relation to group allocation and the outcome assessor will be blind too in relation to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- diet therapy (control) (Active Comparator): Control group undergoing a low calorie diet will not receive supervised pelvic floor muscle training. This group will be assessed at baseline and after 12 weeks. For ethics reason at the end of the study women of the control group will be invited to receive the pelvic floor muscle training program. However, this will not be part of the study.
  Interventions: Other: Pelvic Floor Muscle Training
- Grupo 2 - low calorie diet + PFMT (experimental) (Experimental): The experimental group will receive supervised pelvic floor muscle training in addition to a hypocaloric diet. Women will be instructed to perform daily pelvic floor muscle training at home. 4 sets of 10 maximal voluntary pelvic floor contractions sustained for 6 seconds, followed by 5 voluntary contractions of the pelvic floor muscles. The 4 sets will be performed in 2 different positions (sitting and standing). Once a month, they will receive a supervised in-person session using the same protocol described above, in the other weeks of the month will receive a session supervised by telephysiotherapy once a week. In addition to supervised sessions, women will be encouraged to perform the protocol three more days a week. In addition, they will be instructed to perform "the knack" maneuver.
  Interventions: Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — 4 sets of 10 maximal perceived voluntary pelvic floor contractions sustained for 6 seconds, followed by 5 voluntary pelvic floor muscle contractions. The supervised 4 sets will be performed in 2 different positions (sitting and standing).

SUMMARY:
The purpose of this study is to assess the efficacy of pelvic floor muscle training (PFMT) on urinary incontinence reports in obese women undergoing a low calorie diet prior to bariatric surgery for obesity. The study will also assess and compare rates of adherence to treatments, pelvic floor muscle function and women´s self perception of their PFM function, and satisfaction with treatment.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), the adult overweight rate in 2014 reached 20%, with the highest prevalence among women. In addition to metabolic diseases, obesity can cause musculoskeletal disorders, including pelvic floor muscle (PFM) disorders and urinary incontinence (UI) is the most prevalent one. Conservative intervention can be medication, lifestyle changes, but pelvic floor muscle training (PFMT) is considered the first-line conservative therapy for urinary incontinence in women and it is effective when delivered both individually or in group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the outpatient bariatric surgery service that will start a low calorie diet program as part of the bariatric presurgery routine of the service
* Women
* Over 18 years old
* With body mass index greater than 30kg / m2
* Who have reported urinary incontinence in the last four weeks
* Who have the ability to contract the pelvic floor muscles
* No report of neurological disease, no cognitive impairment
* That are not pregnant.

Exclusion Criteria:

* Women who do not wish to continue participating in the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-08-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
Self report of urinary incontinence by women | Women will be evaluated at baseline
  Self report of urinary incontinence measured using question 3 of the ICIQ-SF. Women will be considered incontinent if they choose option 1,2,3,4,5 of question 3. Women will be considered continent if they choose option 0 of question 3.
Severity and impact of Urinary incontinence in women´s quality of life | Women will be evaluated at baseline
  the severity and impact of Urinary incontinence in women´s quality of life will be measured using the ICIQ-SF score

SECONDARY OUTCOMES:
Participants' adherence to the PFMT protocol | Women will be evaluated at baseline and right after 12 weeks
  Will be assessed using an exercise diary and the complier average causal effects (CACE) method
PFM function | Women will be evaluated at baseline
  the modified Oxford grading scale- MOS (digital vaginal palpation)
participants self-perception of their PFM function | Women will be evaluated at baseline
  women´s self-perception of their PFM function according to the MOS categories
Satisfaction with treatment | only after 12 weeks from the baseline assessment
  Analogic visual scale where 0 represents no satisfaction with treatment and 10 the maximum satisfaction
Subjective satisfaction with treatment | only after 12 weeks from the baseline assessment
  Women will answer the following questions: are you satisfied with the treatment you received for UI? would you do this treatment again ? would you recomend this treatment ? to other people, would you chase another treatment ?
Identification of barriers for the treatment | only after 12 weeks from the baseline assessment
  Women will answer the following questions: Do identifie any barrier or difficulty to adhere to the treatment you received for urinary incontinence?

CONTACTS AND LOCATIONS:
Locations (1):
- Pauliana Carolina de Souza Mendes, Franca, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mendes PCS, Fretta TB, Camargo MFC, Driusso P, Homsi Jorge C. Effect of pelvic floor muscle training on reports of urinary incontinence in obese women undergoing a low-calorie diet before bariatric surgery - protocol of a randomized controlled trial. Trials. 2023 Jun 5;24(1):376. doi: 10.1186/s13063-023-07347-4. PMID 37277833